CLINICAL TRIAL: NCT04496648
Title: The Danish Randomized Sham-Controlled Study of Invasive Versus Medical Treatment for Stable Angina Pectoris
Brief Title: Percutaneous Coronary Intervention Versus Medical Treatment for Stable Angina Pectoris
Acronym: DANANGINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Sune Ammentorp Haahr-Pedersen, Primary Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-18009651
Record Dates: First submitted 2020-06-15; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Coronary Heart Disease; Stable Angina; Ischemic Heart Disease
Keywords: Atherosclerosis; Fractional flow reserve; Optimal medical therapy; Antianginal; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Disease; Angina, Stable; Myocardial Ischemia; Atherosclerosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Randomized patient-blind sham-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Coronary Intervention (Active Comparator): Conventional PCI and optimal medical therapy
  Interventions: Procedure: Percutaneous Coronary Intervention
- Sham-percutaneous coronary intervention (Placebo Comparator): Sham-PCI and optimal medical therapy
  Interventions: Procedure: Sham-percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention with drug-eluting stents and modern techniques
  Other Names: PCI
  Arms: Percutaneous Coronary Intervention
Procedure: Sham-percutaneous coronary intervention — Sham-PCI procedure for at least 15 minutes that includes shifting the C-arm, reinserting the FFR-wire in the catheter and inflating the device.
  Other Names: sham-PCI
  Arms: Sham-percutaneous coronary intervention

SUMMARY:
Patients with ischemic heart disease and symptoms due to lack of oxygen to the heart on exertion (stable angina pectoris) are usually treated by either percutaneous coronary intervention (PCI) or optimal medical therapy (OMT) alone. In patients with mild to moderate coronary artery disease the prognostic impact of PCI is probably limited. Furthermore it is unclear which treatment is superior in terms of relieving symptoms (PCI or OMT). In this trial, patients with mild to moderate coronary artery disease will be randomized to PCI or sham-PCI. All patients will undergo optimal medical therapy. It is hypothesized that PCI is superior to sham-PCI in patients with stable angina pectoris undergoing optimal medical therapy in terms of symptom-relief.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) is a major cause of death and disability worldwide. Patients with ischemic heart disease and symptoms due to lack of oxygen to the heart on exertion (stable angina pectoris) are usually treated by either percutaneous coronary intervention (PCI) or optimal medical therapy (OMT) alone. In patients with mild to moderate coronary artery disease the prognostic impact of PCI is probably limited. Furthermore it is unclear which treatment is superior in terms of relieving symptoms (PCI or OMT). Both treatments are effective in terms of reducing symptoms, but come with potential side effects.

PCI has in previous trials failed to show superiority compared to medical therapy in patients with stable angina pectoris. However, many visually significant lesions do not limit the blood flow significantly to the heart, and stenting such a lesion only exposes the patient to the risk of side effects of intervention. In recent years it has therefore become guideline-recommended practice to perform physiological test to evaluate a potential stenosis. During an angiography this is most often done using fractional flow reserve (FFR).

This study tests the optimal strategy for treatment of angina-symptoms in patients with stable pectoris. PCI is performed with modern stent designs and use of intravascular functional testing (FFR-guided PCI) and compared to sham-PCI.

ELIGIBILITY:
Inclusion criteria

* Age 18-85 years
* Patients with stable angina pectoris undergoing elective coronary angiography
* Canadian Cardiovascular Society (CCS) class 2 or 3
* Informed consent
* Lesions in one or more coronary vessels with a diameter >2.5 mm with FFR-values ≤0.80, and suitable for complete revascularization with PCI.

Exclusion criteria

* Contraindication to PCI or dual antiplatelet therapy (DAPT)
* Use of or indication for oral anticoagulants (OAC) or novel oral anticoagulants (NOAC)
* Use of clopidogrel
* Life expectancy of less than 2 years
* Severe valvular disease
* Severe comorbidity
* Acute coronary event within the past 12 months
* Left ventricular ejection fraction ≤35%.
* Renal function with estimated glomerular filtration rate (eGFR) <30 mL/min
* Pregnant or nursing
* Severe coronary artery disease (left main stenosis, 3-vessel disease, proximal left anterior descending stenosis, chronic total occlusion of major vessel)
* Coronary disease where complete revascularization by PCI is considered difficult or impossible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of strategy success | 3 months
  Number of patients without angina (freedom from angina) and without hospital admission for intolerable stable angina pectoris, unstable angina pectoris, or acute myocardial infarction

SECONDARY OUTCOMES:
Number of all-cause death, any myocardial infarction, stroke, major bleeding, and severe drug reaction | 3 months
  see above
Number of conversions to PCI for procedural complication (sham-PCI group) | 3 months
  see above
Number of patients with hospital admission for intolerable stable angina, unstable angina pectoris, or acute myocardial infarction | 3 months
  see above
Number of patients in CCS class 1, 2, and 3, respectively, without hospital admission for intolerable stable angina, unstable angina pectoris, or acute myocardial infarction | 3 months
  see above
Number of patients with clinically driven coronary revascularization | 3 months
  see above
Change in CCS class | 3 months
  see above
Use of antianginal agents | 3 months
  0, 1, 2, or 3 agents
Quality of life score | 3 months
  5- level EQ-5D (EQ-5D-5L) questionnaire. Each dimension will be scored from 0-5 where a higher score means a better outcome. .
Change in angina-specific quality of life | 3 months
  Seattle Angina Questionnaire 7. Values will range from 0-100 where higher score means better outcome.
Primary composite endpoint in the modified intention-to-treat population | 3 months
  The modified intention-to-treat population is comprised of patients who underwent the study procedure and follow-up without overt or formal unblinding.
Change in CCS class in the modified intention-to-treat population | 3 months
  The modified intention-to-treat population is comprised of patients who underwent the study procedure and follow-up without overt or formal unblinding.
Change in Seattle Angina Questionnaire 7 score in the modified intention-to-treat population | 3 months
  The modified intention-to-treat population is comprised of patients who underwent the study procedure and follow-up without overt or formal unblinding. Values will range from 0-100 where higher score means better outcome.
Change in generic quality of life (EQ-5D-5L) in the modified intention-to-treat population | 3 months
  The modified intention-to-treat population is comprised of patients who underwent the study procedure and follow-up without overt or formal unblinding. Each dimension will be scored from 0-5 where a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Havndrup, Principal Investigator — Zealand Unviersity Hospital; Ole Ahlehoff, Principal Investigator — Odense University Hospital; Ashkan Eftekhari, Principal Investigator — Aarhus University Hospital Skejby; Martin Kirk, Principal Investigator — Aalborg University Hospital; Rikke Sørensen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Gentofte University Hospital, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after publication
Access Criteria: Upon request